CLINICAL TRIAL: NCT03820401
Title: Quantification of Dialysis Performance of Different Dialyzer Membranes With Different Coagulation Strategies, Using a Reference microCT Scanning Technique
Brief Title: Dialysis Performance of Different Dialyzer Membranes Using Different Coagulation Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UGent_FiberClotting_1
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Hemodialysis; Coagulation
Keywords: hemodialyzer; fibre clotting
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Solacea_postHDF_1/1anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro, Japan)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: standard anticoagulation dose
  measurements:
  * blood & dialysate sampling at 60min after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_postHDF_1/2anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: the patient receives only half of his/her standard anticoagulation dose
  measurements:
  * blood & dialysate sampling at 60min after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- FX800_postHDF_1/1anticoagulation (Experimental): intervention:
  * choice of dialyzer: FX800 dialyzer (Fresenius Medical Care, Germany)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: standard anticoagulation dose
  measurements:
  * blood & dialysate sampling at 60min after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- FX800_postHDF_1/2anticoagulation (Experimental): intervention:
  * choice of dialyzer: FX800 dialyzer (Fresenius Medical Care, Germany)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: the patient receives only half of his/her standard anticoagulation dose
  measurements:
  * blood & dialysate sampling at 60min after dialysis start
  * microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_HD_1/1anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro, Japan)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: standard anticoagulation dose
  measurement:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_HD_1/2anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro, Japan)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: the patient receives only half of his/her standard anticoagulation dose
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- FX800_HD_1/1anticoagulation (Experimental): intervention:
  * choice of dialyzer: FX800 dialyzer (Fresenius Medical Care, Germany)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: standard anticoagulation dose
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- FX800_HD_1/2anticoagulation (Experimental): intervention:
  * choice of dialyzer: FX800 dialyzer (Fresenius Medical Care, Germany)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: the patient receives only half of his/her standard anticoagulation dose
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy; Other: preparation of dialyzer
- FX800_HD_1/2anticoagulation_albuprime (Experimental): intervention:
  * choice of dialyzer: FX800 dialyzer (Fresenius Medical Care, Germany)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: the patient receives only half of his/her standard anticoagulation dose
  * preparation of dialyzer: the dialyzer was preprimed with albumin solution
  measurement:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy; Other: preparation of dialyzer
- Evodial_HD_no anticoagulation (Experimental): intervention:
  * choice of dialyzer: Evodial 1.3 (Baxter, USA)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: no anticoagulation is administered
  measurement:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Evodial_HD_no anticoagulation_albuprime (Experimental): intervention:
  * choice of dialyzer: Evodial 1.3 (Baxter, USA)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: no anticoagulation is administered
  * preparation of dialyzer: the dialyzer was preprimed with albumin solution
  measurement:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy; Other: preparation of dialyzer
- Solacea_preHDF_1/4anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: pre dilution hemodiafiltration
  * choice of anticoagulation strategy: the patient receives only 1/4th of his/her standard anticoagulation dose
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_postHDF_1/4anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: the patient receives only 1/4th of his/her standard anticoagulation dose
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_HD_1/4anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: the patient receives only 1/4th of his/her standard anticoagulation dose
  measurements:microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_preHDF_no anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: pre dilution hemodiafiltration
  * choice of anticoagulation strategy: no anticoagulation is administered
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_postHDF_no anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: post dilution hemodiafiltration
  * choice of anticoagulation strategy: no anticoagulation is administered
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy
- Solacea_HD_no anticoagulation (Experimental): intervention:
  * choice of dialyzer: Solacea dialyzer (Nipro Japan)
  * choice of dialysis mode: hemodialysis
  * choice of anticoagulation strategy: no anticoagulation is administered
  measurements:
  - microCT scanning of rinsed and dried dialyzer, post dialysis in order to count open fibers
  Interventions: Device: choice of dialyzer; Other: choice of dialysis mode; Other: choice of anticoagulation strategy

INTERVENTIONS:
Device: choice of dialyzer — Fiber blocking is calculated in different commercially available dialyzers
Other: choice of dialysis mode — Fiber blocking is calculated in different commercially available dialyzers used in different dialysis stategies
Other: choice of anticoagulation strategy — Fiber blocking is calculated in different commercially available dialyzers using different anticoagulation strategies
Other: preparation of dialyzer — Fiber blocking is calculated in different commercially available dialyzers either preprimed with Albumin or not
  Arms: Evodial_HD_no anticoagulation_albuprime; FX800_HD_1/2anticoagulation; FX800_HD_1/2anticoagulation_albuprime

SUMMARY:
Coagulation within the dialyzer membrane fibres is an obvious biological sign of bio-incompatibility. To avoid clotting during extracorporeal treatment, an anticoagulant is added to the circuit, resulting in an increased risk for bleeding complications.

In addition, there is evidence that a substantial number of fibers can become blocked before this is reflected in routinely observed parameters, or in termination of the dialysis session. Little is known about the impact of such subclinical clotting on dialyzer performance in terms of solute clearance.

Membrane clogging due to deposition of proteins and red blood cells on the dialysis membrane may influence both the diffusive and convective transport characteristics of the dialyzer membrane before leading to complete dialyzer clotting.

In 2018, the invesitgators described a method to objectively count the number of blocked fibres inside a dialyzer using a micro-CT scanning technique.

In the present trial, the investigators use this method to assess the resistance of the dialyzer to clotting, and to evaluate the impact of subclinical fibre blocking on solute removal and thus performance of a dialyzer during a dialysis session.

The aim of this randomized cross-over study is to objectively quantify the performance of different dialyzer membranes: ATA™ membrane in the Solacea™ dialyzer, polysulfone membrane in the FX800 dialyzer, and the heparin-coated AN membrane in the Evodial dialyzer, and this with different anticoagulation strategies.

DETAILED DESCRIPTION:
This single centre, randomized cross-over study includes ten consecutive stable chronic hemodialysis (HD) patients who experienced stable dialysis sessions during the last 4 weeks, and had no known coagulation disorder, active inflammation or malignancy.

Double-needle vascular access is achieved through a native arterio-venous fistula or a well-functioning double lumen tunnelled central venous catheter.

In a first test series, each patient is dialyzed for 240min (at midweek) in 4 different regimens, randomly using 2 different dialyzers and 2 different anticoagulation schemes. Patients receive their regular brand of Low-Molecular-Weight Heparin anticoagulation at the beginning of the dialysis session, and this randomly either at their regular dose (full dose 1/1) or at only 50% of their regular dose (half dose 1/2). All test sessions are performed with blood flow at 300mL/min and dialysate flow at 500mL/min in post dilution hemodiafiltration (HDF) mode (substitution flow 75mL/min). Ultrafiltration rates is set according to the patient's interdialytic weight gain and clinical status:

1. ATA™ Solacea 19H - HDF - 1/1 anticoagulation
2. ATA™ Solacea 19H - HDF - 1/2 anticoagulation
3. polysulfone FX800 - HDF - 1/1 anticoagulation
4. polysulfone FX800 - HDF - 1/2 anticoagulation

During the 4 experimental midweek sessions, blood is sampled from the arterial and venous blood lines, and spent dialysate is sampled from the outlet line, all at 60min after the dialysis start. Blood samples are immediately centrifuged and serum and dialysate are stored at -80°C until batch analysis.

Concentrations of urea, kappa and lambda free light chains, and myoglobin are determined. Extraction ratios and adsorption on the membrane are calculated from concentrations.

At the end of the dialysis session, a standard rinsing procedure of the hemodialyzer is performed using exact 300mL rinsing solution. Next, the hemodialyzer is dried using continuous positive pressure ventilation. Dialyzer fibre blocking is visualized in the dialyzer outlet potting using a 3D CT scanning technique on micrometer resolution. HECTOR is a High Energy CT scanner Optimized for Research, built by the Ghent University Centre for X-ray Tomography (UGCT) in collaboration with the UGCT spin-off company XRE (Gent, Belgium). In front of the X-ray source, the dialyzer is mounted vertically on a precision rotation stage, and radiographies were recorded over 360° with an angular interval of 0.15°. Scan conditions are optimized to maximize the signal-to-noise ratio based on the sample size and structure, and the scanner properties. The tube voltage is set at 80kV, at a power of 20 Watts, the maximal power that allowed imaging at a resolution of 25µm. A total of 2401 projections are recorded with 500ms exposure each, resulting in a total exposure time of 20 minutes. Acquired images at 0 (projection 1) and 360° (projection 2401) are compared to exclude movement of the hemodialyzer during the scanning process. Reconstruction of the raw projection data is performed with the Octopus Reconstruction software package, licensed by XRE23.

Fibers are counted in the central cross-section of the dialyzer outlet potting in a computer-based way using the Fiji image processing toolkit of ImageJ analysis software (ImageJ 1.51H, NIH, Bethesda, USA), an open-source platform for biological-image analysis.

In a second test series in 10 stable HD patients, no blood sampling is performed but dialyzers are scanned post dialysis. The following different dialyzers in HD modus at midweek are tested:

1. ATA™ Solacea 19H - HD - 1/1 anticoagulation
2. ATA™ Solacea 19H - HD - 1/2 anticoagulation
3. polysulfone FX800 - HD - 1/1 anticoagulation
4. polysulfone FX800 - HD - 1/2 anticoagulation
5. polysulfone FX800 - HD - 1/2 anticoagulation - with predialysis albmuin priming of the membrane
6. Evodial - HD - no anticoagulation
7. Evodial - HD - no anticoagulation - with predialysis albmuin priming of the membrane

In a third test series in 10 stable HD patients, no blood sampling is performed but dialyzers are scanned post dialysis. The following different dialyzers at midweek are tested:

1. ATA™ Solacea 19H - pre dilution HDF (substitution 150mL/min) - 1/4 anticoagulation
2. ATA™ Solacea 19H - post dilution HDF (substitution 75mL/min) - 1/4 anticoagulation
3. ATA™ Solacea 19H - HD - 1/4 anticoagulation
4. ATA™ Solacea 19H - pre dilution HDF (substitution 150mL/min) - no anticoagulation
5. ATA™ Solacea 19H - post dilution HDF (substitution 75mL/min) - no anticoagulation
6. ATA™ Solacea 19H - HD - no anticoagulation

First outcome measure: relative number of open fibers in each tested dialyzer. Second outcome measure: dialyzer performance (extraction ratio, adsorption).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* experienced stable dialysis sessions during the last 4 weeks
* double needle/lumen well-functioning vascular access

Exclusion Criteria:

* known coagulation disorder
* active inflammation
* malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Number of open fibres in the dialyzer | 17 weeks
  Number of open fibres as assessed post dialysis by a reference microCT scanning technique

SECONDARY OUTCOMES:
Extraction ratio of three middle molecules in the dialyzer | 4 weeks
  Extraction ratio from myoglobin, kappa and lambda free light chains as calculated from their concentrations at the dialyzer inlet en outlet

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital - Nephrology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vanommeslaeghe F, Van Biesen W, Dierick M, Boone M, Dhondt A, Eloot S. Micro-computed tomography for the quantification of blocked fibers in hemodialyzers. Sci Rep. 2018 Feb 8;8(1):2677. doi: 10.1038/s41598-018-20898-w. PMID 29422614
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593